CLINICAL TRIAL: NCT06297915
Title: Evaluation and Comparison of the Effectiveness of Ketamine and Lidocaine Infusion in Peripheral Neuropathic Pain: A Retrospective Study
Brief Title: Infusion Treatments of Chronic Peripheral Neuropathic Pain
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Tugce Yavuz, Medical Doctor, Hacettepe University
Other Study IDs: 2022/08-45
Record Dates: First submitted 2024-03-01; First posted 2024-03-07 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Neuropathic Pain
Keywords: Lidocaine; Ketamine; Pain measurement, scale
MeSH Terms: conditions — Neuralgia | interventions — Ketamine

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Ketamine — Ketamine infusion was administered at 1 mg/kg (in 1 hour)
  Other Names: Group K
Drug: Lidocain — Lidocaine infusion was administered at 3 mg/kg (in 1 hour)
  Other Names: Group L

SUMMARY:
This study aimed to evaluate and compare the efficacy of ketamine and lidocaine infusion in patients with chronic peripheral neuropathic pain.

Patients who received intravenous ketamine infusion and the other patient group who received intravenous lidocaine infusion were evaluated in the study. Pain scores and quality of life were assessed with scales before treatment at two weeks, two months, and six months after treatment.

DETAILED DESCRIPTION:
This study, it was aimed to evaluate and compare the efficacy of intravenous infusion of ketamine and lidocaine, which have been known and used in pain management and which have recently increased interest in the treatment of peripheric neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* Patients with peripheral neuropathic pain (radicular neuropathy, diabetic neuropathy, complex regional pain syndrome type 2, traumatic peripheral nerve injury, trigeminal neuralgia, postherpetic neuralgia)
* Patients who was evaluated by DN4 scores with of ≥4 points

Exclusion Criteria:

* Patients with central nervous system disease .
* Patients with cancer related neuropatic pain.
* Patients with central neuropathic pain patterns.
* Patients with renal, hepatic, cardiovascular, and psychiatric diseases.
* Patients whose treatment could not be completed due to side effects or other reasons.
* Patients who had lost their follow-up .

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: For the retrospectively designed study, data (electronic database program of the hospital and files) of the patients admitted to the algology clinic with neuropathic pain symptoms between January 2021 and May 2021 were evaluated.
Sampling Method: Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2022-05-17 (Actual); Primary Completion 2023-05-10 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Neuropathic Pain Scale | Before treatment at two weeks, two months, and six months after treatment.The 7 symptoms items are scored by interviewing the patient.The scores are added and a score of 4 or more outout of ,10 point (severe pain ) is suggestive of neuropathic pain.
  Neuropathic Pain 4 Questions (DN4)
Pain Rating Scale | Before treatment at two weeks, two months, and six months after treatment.NRS in which individuals rate their pain on an ten-point numerical scale. Zero:''no pain at all' ten-point ''severe pain''
  Numeric Rating Scale

SECONDARY OUTCOMES:
Quality of Life Scale | Before treatment at two weeks, two months, and six months after treatment.12-question survey PCS and the MCS Scores above 50 indicate a better-than-average health-related quality of life, while scores below 50 suggest below-average health.
  Short form-12 (SF-12)

CONTACTS AND LOCATIONS:
Overall Officials: Gokhan Sucu, MD, Study Chair — HACETTEPE UNIVERSİTY
Locations (1):
- Hacettepe University, Ankara, Cankaya, Turkey (Türkiye)

REFERENCES:
- [Background] Niesters M, Martini C, Dahan A. Ketamine for chronic pain: risks and benefits. Br J Clin Pharmacol. 2014 Feb;77(2):357-67. doi: 10.1111/bcp.12094. PMID 23432384
- [Background] van der Wal SE, van den Heuvel SA, Radema SA, van Berkum BF, Vaneker M, Steegers MA, Scheffer GJ, Vissers KC. The in vitro mechanisms and in vivo efficacy of intravenous lidocaine on the neuroinflammatory response in acute and chronic pain. Eur J Pain. 2016 May;20(5):655-74. doi: 10.1002/ejp.794. Epub 2015 Dec 18. PMID 26684648
- [Background] Shteamer JW, Callaway MA, Patel P, Singh V. How effective is ketamine in the management of chronic neuropathic pain? Pain Manag. 2019 Nov;9(6):517-519. doi: 10.2217/pmt-2019-0032. Epub 2019 Oct 15. No abstract available. PMID 31613180
- [Background] Jendoubi A, Naceur IB, Bouzouita A, Trifa M, Ghedira S, Chebil M, Houissa M. A comparison between intravenous lidocaine and ketamine on acute and chronic pain after open nephrectomy: A prospective, double-blind, randomized, placebo-controlled study. Saudi J Anaesth. 2017 Apr-Jun;11(2):177-184. doi: 10.4103/1658-354X.203027. PMID 28442956